CLINICAL TRIAL: NCT06819839
Title: Impact of a Community Health Worker Care Model to Reduce Cardiovascular Disease Risk Among Conflict-affected Populations in Eastern Myanmar: a Cluster Randomized Controlled Trial (cRCT)
Brief Title: Community-led Strategy to Reduce Cardiovascular Disease Risk Among Conflict-affected Populations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Community Partners International (Other)
Collaborators: Khon Kaen University (Other); George Washington University (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NCR245957
Record Dates: First submitted 2025-01-25; First posted 2025-02-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases; Hypertension; Diabetes
Keywords: Cardiovascular disease (CVD); Village health worker; Eastern Myanmar; Hypertension; Diabetes; Care delivery model
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Diabetes Mellitus | interventions — Community Health Workers

STUDY DESIGN:
Intervention Model Description: Cluster Randomized Controlled Trial in 13 villages
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Village Health Worker (VHW) Care Model (Experimental): 7 villages are randomly selected and people (40 years and above) with increased cardiovascular disease risk receive VHW Care
  Interventions: Behavioral: Village Health Worker (VHW) Care Model
- Standard Community Care (No Intervention): 6 control villages randomly selected from 6 matched pairs and triplets of villages, and conduct a baseline and endline survey

INTERVENTIONS:
Behavioral: Village Health Worker (VHW) Care Model — VHW care model includes four components: (1) universal screening of all non-pregnant adults over 40 for elevated CVD risk (2) confirmatory visit to confirm diagnoses of hypertension, diabetes and elevated CVD risk (predicted 10-year risk >10%) (3) monthly household visits by VHW; (4) an mHealth tool (tablet computer) to assist with determination of study eligibility and provide recommendations for initiation of medications according to local guidelines. VHW household visits include: health education on smoking cessation, healthy diet, physical activity and medication adherence; assessment of possible medication side effects, measurement of blood pressure and (when applicable) blood glucose; review monitoring results with the treating clinician household delivery of medications; and facilitate referral and transport to higher levels of care.
  Arms: Village Health Worker (VHW) Care Model

SUMMARY:
The goal of this study is to test a village health worker (VHW) based care model to reduce cardiovascular risk among adults in areas of eastern Myanmar affected by armed conflict. All individuals aged 40 years and above will be invited to participate in this study. Participants will be checked whether they have a history of cardiovascular disease, diabetes (high blood sugar), high blood pressure or risk of developing cardiovascular disease by asking for medical history, measuring blood pressure, weight and height, and blood glucose if necessary. The main question the study aims to answer is:

Does villagers residing in the VHW supported villages have their blood pressure controlled, adherent to therapy and subsequently reduce the risk of developing cardiovascular disease after 5 months of monthly VHW home visits?

DETAILED DESCRIPTION:
Myanmar is a Southeast Asian country which has been struggling with active conflict situation since 2021 - resulting massive internal displacement especially in ethnic areas. It is widely known that Community- and village-health worker (VHW) led interventions have reduced CVD risk in stable areas of low and middle income countries, but have not been adapted for internally displaced people (IDPs) exposed to active conflict. In addition, CVD is the leading cause of death in Myanmar and according to recent national survey, 75% of adults have at least one CVD risk factor.

This cRCT study is a third phase of the "Implementation of a community-led strategy to reduce cardiovascular disease risk among conflict-affected populations in eastern Myanmar" and Phase 1 and 2 have been successfully completed. The VHW care model was developed based on a Causal Loop Analysis (CLA) workshop in Phase 1 (GWU IRB# NCR234977), which included a Qualitative Study, Causal Loop Analysis workshop and Village Health Worker Intervention Design. The VHW care model was then tested in the Phase 2 Feasibility study (GWU IRB # NCR235114) in 3 villages conducted over three months (November 2023-January 2024).

Specific aim of this study includes:

1. to assess the impact of a village health worker (VHW) care model in reducing cardiovascular disease (CVD) risk in rural Myanmar by conducting a cluster randomized trial in 13 villages surrounding 3 clinics.

   Hypothesis: High proportions of villagers over 40 are screened for elevated CVD risk (>90%), attend a confirmatory visit (>85%), initiate a high proportion of evidence-based therapies (>75%), participate in at least one follow-up visit (>70%) and are adherent to therapy at three months (>50%).
2. to evaluate implementation of the VHW CVD program using the REAIM-PRISM framework.

   Hypothesis: The VHW CVD intervention has broad reach, is acceptable, effective, is widely adopted, and perceived to be sustainable by community partners.
3. to establish the time and cost required to carry out VHW care model activities as well as their impact on the care cascade for CVD risk, from screening to linkage to care, initiation of therapy and retention in care.

Hypothesis: The VHW CVD intervention is cost-effective, affordable, and sustainable.

Advantage of the study:

The VHW care model extends basic monitoring and treatment functions for chronic disease management to remote rural villages where physical terrain, high transportation cost and insecurity limit options for transportation to and from centralized clinic locations. Via VHWs, patient medication adherence, blood pressure, and blood glucose (when relevant) will be reported to treating clinicians (medics). Medics will be able to use this information to either schedule an in-person visit or to remotely refill or titrate medications.

ELIGIBILITY:
Inclusion criteria

* Aged 40 years or older
* Current resident of study villages
* No previous history of screening during the feasibility study a year ago
* At least one CVD risk factor

Exclusion criteria

- Currently pregnant or within three months postpartum

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2024-10-27 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence - self-reported MARS-5 | 5 months
  Proportion of individuals adherent to evidence-based medications (taking the medication within the past 2 weeks, from self-report), AND a medication adherence report scale (MARS-5) adherence score of at least 16 out of 25. Requires taking at least one medication from each of the classes for which the individual is eligible: anti-hypertensive medication for individuals with hypertension, and statin for individuals with a history of ischemic heart disease, history of stroke, diabetes or 10-year CVD risk >10%.

SECONDARY OUTCOMES:
Change in medication adherence - self reported high | 5 months
  Proportion of individuals with high self reported adherence to evidence-based medications for which they are eligible. Requires taking at least one medication from each of the classes for which the individual is eligible (see primary outcome), AND a MARS-5 adherence scale of at least 20 out of 25. The MARS-5 adherence scale has a range from 5 to 25, with higher scores representing higher self-reported adherence.
Change in medication adherence - lenient | 5 months
  Proportion of individual taking at least one among any of the evidence-based medication classes s/he is eligible for (less strict definition medication adherence)
Change in population level adherence | 5 months
  Population level adherence, calculated as the ratio of the sum of the medication classes taken divided by the sum of eligible medication classes, among all individuals in the group. For example, if individual 1 is eligible for and takes one medication and if individual is eligible for two medications but takes only one, then population level adherence = (1+1) / (1+ 2) = 0.66.
Change in adherence to blood pressure medication | 5 months
  Respective proportions reporting 'moderate' or 'high' adherence to blood pressure medications using 'low' (5 to 15), 'moderate' (16 to 20) or 'high' (21-25) on the MARS-5 adherence scale. The MARS-5 adherence scale has a range from 5 to 25, with higher scores representing higher self-reported adherence.
Change in adherence to statin medication | 5 months
  Respective proportions reporting 'low', 'moderate' or 'high' adherence to blood pressure medications using 'low' (5 to 15), 'moderate' (16 to 20) or 'high' (21-25 on the MARS-5 adherence scale. The MARS-5 adherence scale has a range from 5 to 25, with higher scores representing higher self-reported adherence.
Change in mean MARS-5 adherence score | 5 months
  Among individuals eligible for either blood pressure or statin medication. The MARS-5 adherence scale has a range from 5 to 25, , with higher scores representing higher self-reported adherence.
Change in first and recurrent CVD event risk | 5 months
  Change in CVD event risk is assessed using a modified relative risk reduction tool that accurately quantifies longitudinal changes in cardiovascular disease risk.
Change in mean CVD risk predicted by World Health Organization CVD risk calculator | 5 months
  Change in mean CVD risk is the difference between the mean 10-year CVD risk of participants eligible for treatment at endline and the mean 10-year CVD risk of eligible individuals at baseline, as calculated using the WHO CVD risk equation. This method is known to inaccurately estimate change in CVD risk; it is reported for the sake of comparison to studies that (mis)use the WHO risk equation to define outcomes.
Change in relative Go Score | 5 months
  The relative GO score is defined as the proportion of benefit (relative CVD risk reduction) achieved, out of the maximum benefit possible from guideline directed therapy. The two therapies in the current study are blood pressure medications and statins. The GO Score has minimum value of zero and maximum value of one, with higher values representing a better outcome (greater proportion of possible benefit achieved). The relative GO Score is calculated using the ratio of relative risk reduction achieved divided by the relative risk reduction possible.
Change in absolute Go Score | 5 months
  The absolute GO score is defined as the proportion of absolute benefit (absolute CVD risk reduction) achieved, out of the maximum benefit possible from guideline directed therapy. The two therapies in the current study are blood pressure medications and statins. The GO Score has minimum value of zero and maximum value of one, with higher values representing a better outcome (greater proportion of possible benefit achieved). The absolute GO Score is calculated using the ratio of absolute risk reduction achieved to the absolute risk reduction possible.
Care cascade step 1: proportion aware of their diagnosis | 5 months
  Proportion of the number of participants aware of their diagnoses (hypertension, diabetes and elevated CVD risk) to adults over 40 years eligible for statins, anti-hypertensive treatment, or both statins and anti-hypertensives
Care cascade step 2: proportion linked to care | 5 months
  Proportion of participants linked to care (at least 1 clinic visit or VHW visit for CVD risk management) among adults over 40 years eligible for treatment
Care cascade step 3: proportion initiated on appropriate medications | 5 months
  Proportion of participants initiated on appropriate medications among adults over 40 years eligible for treatment.
Care cascade step 4: proportion taking appropriate medication | 5 months
  Proportion of participants who report taking appropriate medication in the past two weeks among adults over 40 years eligible for treatment
Care cascade step 5: proportion adherent to treatment | 5 months
  Proportion of participants who report taking appropriate medication in the past two weeks AND who report adherence to treatment, where adherence is defined as 16-25 on the MARS-5 adherence scale. The MARS-5 adherence scale has a range from 5 to 25, , with higher scores representing higher self-reported adherence.
Hypertension Care cascade step 1: proportion aware of their diagnosis | 5 months
  Proportion of the number of participants aware of their diagnoses (hypertension, diabetes and elevated CVD risk) to adults over 40 years eligible for statins, anti-hypertensive treatment, or both statins and anti-hypertensives
Hypertension Care cascade step 2: proportion linked to care | 5 months
  Proportion of participants linked to care (at least 1 clinic visit or VHW visit for CVD risk management) among adults over 40 years eligible for treatment
Hypertension Care cascade step 3: proportion initiated on appropriate medications | 5 months
  Proportion of participants initiated on appropriate medications among adults over 40 years eligible for treatment.
Hypertension Care cascade step 4: proportion taking appropriate medication | 5 months
  Proportion of participants who report taking appropriate medication in the past two weeks among adults over 40 years eligible for treatment
Hypertension Care cascade step 5: proportion adherent to treatment | 5 months
  Proportion of participants who report taking appropriate medication in the past two weeks AND who report adherence to treatment, where adherence is defined as 16-25 on the MARS-5 adherence scale. The MARS-5 adherence scale has a range from 5 to 25, , with higher scores representing higher self-reported adherence.
Hypertension Care cascade step 6: proportion with systolic blood pressure below 140mmHg | 5 months
  Proportion of participants with systolic blood pressure below 140mmHg among adults over 40 years with hypertension
Hypertension Care cascade step 7: proportion with systolic blood pressure below 130mmHg | 5 months
  Proportion of participants with systolic blood pressure below 130mmHg among adults over 40 years with hypertension
Hypertension Care cascade step 8: proportion with systolic blood pressure below 120mmHg | 5 months
  Proportion of participants with systolic blood pressure below 120mmHg among adults over 40 years with hypertension
Statin care cascade step 1: proportion linked to care | 5 months
  Proportion of participants linked to care (at least 1 clinic visit or VHW visit for CVD risk management) among adults over 40 years eligible for statin treatment
Statin care cascade step 2: proportion initiated on appropriate medications | 5 months
  Proportion of participants initiated on appropriate medications among adults over 40 years eligible for treatment.
Statin care cascade step 3: proportion taking appropriate medication | 5 months
  Proportion of participants who report taking appropriate medication in the past two weeks among adults over 40 years eligible for treatment
Statin care cascade step 4: proportion adherent to statin treatment | 5 months
  Proportion of participants who report taking appropriate medication in the past two weeks AND who report adherence to treatment, where adherence is defined as 16-25 on the MARS-5 adherence scale. The MARS-5 adherence scale has a range from 5 to 25, , with higher scores representing higher self-reported adherence.
Change in mean systolic blood pressure in the hypertensive population | 5 months
  Changes in blood pressure is the difference between the mean systolic blood pressure at baseline and the mean systolic blood pressure at endline, among individuals with likely hypertension, defined as taking anti-hypertensive treatment.
Change in current smoking prevalence | 5 months
  Current smoking is assessed by an affirmative answer to the question "In the past two weeks have participant smoked any tobacco products, such as cigarettes, cigars or pipes?", asked on individuals with likely eligible for blood pressure medication or statin treatment. Smoking prevalence is defined as the proportion of current smokers among all adults 40 years or older.
Mean change in systolic blood pressure among individuals with hypertension who have repeated measures | 5 months
  Changes in systolic blood pressure is the (paired) mean difference in systolic blood pressure from baseline to endline change , among individuals with likely hypertension who have measurements at baseline and endline. In intervention villages individuals with repeated measures were assessed during village screening at baseline and the endline assessments; in control villages individuals with repeated measures represent approximately one-quarter of individuals who expected to participate in both baseline and endline household surveys (both surveys target half of all households, hence the probability of being selected at both baseline and endline is approximately 0.25).
Smoking cessation (quit) rate among smokers with repeated measures | 5 months
  Current smoking is assessed by an affirmative answer to the question "In the past two weeks have participant smoked any tobacco products, such as cigarettes, cigars or pipes?", asked of individuals eligible for anti-hypertension or statin treatment. Smoking cessation (quite rate) is defined as the proportion of current smokers at baseline who do not report current smoking at endline. In intervention villages individuals with repeated measures were assessed during village screening at baseline and the endline assessments; in control villages individuals with repeated measures represent approximately one-quarter of individuals who expected to participate in both baseline and endline household surveys (both surveys target half of all households, hence the probability of being selected at both baseline and endline is approximately 0.25).
Change in medication adherence among individuals with repeated measures | 5 months
  Proportion of individuals adherent to evidence-based medications (taking the medication within the past 2 weeks, from self-report), AND a medication adherence report scale (MARS-5) adherence score of at least 16 out of 25. Requires taking at least one medication from each of the classes for which the individual is eligible: anti-hypertensive medication for individuals with hypertension, and statin for individuals with a history of ischemic heart disease, history of stroke, diabetes or 10-year CVD risk >10%. In intervention villages individuals with repeated measures were assessed during village screening at baseline and the endline assessments; in control villages individuals with repeated measures represent approximately one-quarter of individuals who expected to participate in both baseline and endline household surveys (both surveys target half of all households, hence the probability of being selected at both baseline and endline is approximately 0.25).
Changes in GO Score among individuals with repeated measures | 5 months
  Changes in GO Score is the difference between observed changes in blood pressure and smoking cessation among individuals at endline AND observed changes in blood pressure and smoking cessation among individuals at baseline. The GO Score has minimum value of zero and maximum value of one, with higher values representing a better outcome (greater proportion of possible benefit achieved).
Effect modification by presence of a disability | 5 months
  Disability is defined as either "a lot of difficulty" or "cannot do at all" in relation to at least one of 8 disability function items from the Washington Group - Extended Set on Function (WG-ES)
Effect modification by 10-year (predicted) CVD risk | 5 months
  Using 10-year (predicted) CVD risk
Effect modification by Sex | 5 months
  Stratified by male and female
Effect modification by Age | 5 months
  Stratified by age groups (40-49 years, 50-59, 60-69, 70+)
Effect modification by household wealth | 5 months
  Using Myanmar wealth quintiles defined by Equity tool
Effect modification by respondent educational attainment | 5 months
  Using Educational attainment
Effect modification by income | 5 months
  Using level of income
Effect modification by residential status in the village | 5 months
  Residential status is defined as arrival before/after initial screening (dichotomous)
Multidimensional index of vulnerability | 5 months
  The multidimensional index of vulnerability will be calculated as a multivariate propensity score of the primary dichotomous outcome, using the predicted probability from a logistic regression model that includes multiple axes of disadvantage as predictors including household wealth, educational attainment, income, women's empowerment and distance from a health facility. The index has a minimum value of 0 and maximum value of 1. Increasing values represent higher vulnerability.
Changes in relative inequities in primary and secondary outcomes: the relative concentration index | 5 months
  Relative health inequities will be summarized on the relative scale using the relative concentration index, a summary health equity metric developed by the World Bank. The relative concentration index has a range from zero to 1 (though the range for dichotomous outcomes is 'bounded', with a lower maximum value that varies as a function of the proportion of the outcome.
Changes in absolute inequities in primary and secondary outcomes: the absolute concentration index | 5 months
  Absolute health inequities will be summarized on the absolute scale using the absolute concentration index, a summary health equity metric developed by the World Bank, and equal to the mean value in the population multiplied by the relative concentration index (see Wagstaff et al 2002).
Changes in equity-weighted primary and secondary outcomes: the achievement index | 5 months
  We will calculate the achievement index, an equity-weighted health outcome metric developed by the World Bank, and equal to the mean value in the population multiplied by (1 minus the relative concentration index); (see Wagstaff et al 2002).
Linkage to care cascade 1: proportion of adults screened for CVD risk factors | 5 months
  Proportion of population >40 years old who complete screening questionnaire, in intervention villages
Linkage to care cascade 2: proportion of adults who complete a confirmatory visit | 5 months
  Proportion of population >40 years old who complete confirmatory visit, among adults eligible for a confirmatory visit
Linkage to care cascade 3: proportion of adults eligible for the longitudinal study who attended at least one VHW visit | 5 months
  Proportion of adults eligible for the longitudinal study who attended at least one VHW visit
Linkage to care cascade 4: proportion retained in care at the end of the study | 5 months
  Retained in care is defined as not withdrawn from the study participated in a VHW visit in the previous 60 days
Mean number (n, %) of VHW visits completed | 5 months
  Mean number (n, %) of VHW visits completed among eligible population
Mean number (n, %) of medic visits per participant | 5 months
  Mean number (n, %) of medic visits per participant among eligible population
Refused participation, among eligible individuals (n, %) | 5 months
  Number (n, %) of individuals among eligible population who refused to participate in the study
Withdrew from study | 5 months
  Number (n, %) of individuals among eligible population who withdrew from study
Deceased (n, %) | 5 months
  Number (n,%) of individuals among eligible population who died during the duration of the study
Referrals for acute symptoms or other complication | 5 months
  Number (n, %) of individuals among eligible population who received referrals for acute symptoms or other complication
Proportion of visits with adequate quality clinical decision-making | 5 months
  Proportion of visits with adequate quality clinical decision-making from a logbook chart review

CONTACTS AND LOCATIONS:
Overall Officials: Adam Richards, Principal Investigator — George Washington University
Locations (1):
- Community Partners International, Hpa-An, Kayin State, Burma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nagamine Y, Shobugawa Y, Sasaki Y, Takagi D, Fujiwara T, Khin YP, Nozaki I, Shirakura Y, Kay Thi L, Poe Ei Z, Thae Z, Win HH. Associations between socioeconomic status and adherence to hypertension treatment among older adults in urban and rural areas in Myanmar: a cross-sectional study using baseline data from the JAGES in Myanmar prospective cohort study. BMJ Open. 2023 Jan 17;13(1):e065370. doi: 10.1136/bmjopen-2022-065370. PMID 36653052
- [Background] Lloyd-Jones DM, Huffman MD, Karmali KN, Sanghavi DM, Wright JS, Pelser C, Gulati M, Masoudi FA, Goff DC Jr. Estimating Longitudinal Risks and Benefits From Cardiovascular Preventive Therapies Among Medicare Patients: The Million Hearts Longitudinal ASCVD Risk Assessment Tool: A Special Report From the American Heart Association and American College of Cardiology. Circulation. 2017 Mar 28;135(13):e793-e813. doi: 10.1161/CIR.0000000000000467. Epub 2016 Nov 4. PMID 27815375
- [Background] Kaur G, Chauhan AS, Prinja S, Teerawattananon Y, Muniyandi M, Rastogi A, Jyani G, Nagarajan K, Lakshmi P, Gupta A, Selvam JM, Bhansali A, Jain S. Cost-effectiveness of population-based screening for diabetes and hypertension in India: an economic modelling study. Lancet Public Health. 2022 Jan;7(1):e65-e73. doi: 10.1016/S2468-2667(21)00199-7. Epub 2021 Nov 12. PMID 34774219
- [Background] Basu S, Wagner RG, Sewpaul R, Reddy P, Davies J. Implications of scaling up cardiovascular disease treatment in South Africa: a microsimulation and cost-effectiveness analysis. Lancet Glob Health. 2019 Feb;7(2):e270-e280. doi: 10.1016/S2214-109X(18)30450-9. Epub 2018 Dec 6. PMID 30528531
- [Background] Brownell NK, Ziaeian B, Jackson NJ, Richards AK. Trends in Income Inequities in Cardiovascular Health Among US Adults, 1988-2018. Circ Cardiovasc Qual Outcomes. 2024 May;17(5):e010111. doi: 10.1161/CIRCOUTCOMES.123.010111. Epub 2024 Apr 3. PMID 38567505
- [Background] Patel A, Praveen D, Maharani A, Oceandy D, Pilard Q, Kohli MPS, Sujarwoto S, Tampubolon G. Association of Multifaceted Mobile Technology-Enabled Primary Care Intervention With Cardiovascular Disease Risk Management in Rural Indonesia. JAMA Cardiol. 2019 Oct 1;4(10):978-986. doi: 10.1001/jamacardio.2019.2974. PMID 31461123
- [Background] Schwalm JD, McCready T, Lopez-Jaramillo P, Yusoff K, Attaran A, Lamelas P, Camacho PA, Majid F, Bangdiwala SI, Thabane L, Islam S, McKee M, Yusuf S. A community-based comprehensive intervention to reduce cardiovascular risk in hypertension (HOPE 4): a cluster-randomised controlled trial. Lancet. 2019 Oct 5;394(10205):1231-1242. doi: 10.1016/S0140-6736(19)31949-X. Epub 2019 Sep 2. PMID 31488369
- [Background] Jafar TH, Jehan I, de Silva HA, Naheed A, Gandhi M, Assam P, Finkelstein EA, Quigley HL, Bilger M, Khan AH, Clemens JD, Ebrahim S, Turner EL; for COBRA-BPS Study Group; Kasturiratne A. Multicomponent intervention versus usual care for management of hypertension in rural Bangladesh, Pakistan and Sri Lanka: study protocol for a cluster randomized controlled trial. Trials. 2017 Jun 12;18(1):272. doi: 10.1186/s13063-017-2018-0. PMID 28606184
- [Background] Jafar TH, Gandhi M, de Silva HA, Jehan I, Naheed A, Finkelstein EA, Turner EL, Morisky D, Kasturiratne A, Khan AH, Clemens JD, Ebrahim S, Assam PN, Feng L; COBRA-BPS Study Group. A Community-Based Intervention for Managing Hypertension in Rural South Asia. N Engl J Med. 2020 Feb 20;382(8):717-726. doi: 10.1056/NEJMoa1911965. PMID 32074419
- [Background] Patenaude B, Odihi D, Sriudomporn S, Mak J, Watts E, de Broucker G. A standardized approach for measuring multivariate equity in vaccination coverage, cost-of-illness, and health outcomes: Evidence from the Vaccine Economics Research for Sustainability & Equity (VERSE) project. Soc Sci Med. 2022 Jun;302:114979. doi: 10.1016/j.socscimed.2022.114979. Epub 2022 Apr 16. PMID 35462106
- [Background] Chakraborty NM, Fry K, Behl R, Longfield K. Simplified Asset Indices to Measure Wealth and Equity in Health Programs: A Reliability and Validity Analysis Using Survey Data From 16 Countries. Glob Health Sci Pract. 2016 Mar 25;4(1):141-54. doi: 10.9745/GHSP-D-15-00384. Print 2016 Mar. PMID 27016550
- [Background] Eddy DM, Adler J, Morris M. The 'Global Outcomes Score': a quality measure, based on health outcomes, that compares current care to a target level of care. Health Aff (Millwood). 2012 Nov;31(11):2441-50. doi: 10.1377/hlthaff.2011.1274. PMID 23129674
- [Background] Spetz K, Olbers T, Ostbring M, Moon Z, Horne R, Andersson E. Using the 5-Item Medication Adherence Report Scale (MARS-5) to Screen for Non-adherence to Vitamin and Mineral Supplementation After Bariatric Surgery. Obes Surg. 2024 Feb;34(2):576-582. doi: 10.1007/s11695-023-07027-x. Epub 2024 Jan 4. PMID 38177555
- [Background] Chan AHY, Horne R, Hankins M, Chisari C. The Medication Adherence Report Scale: A measurement tool for eliciting patients' reports of nonadherence. Br J Clin Pharmacol. 2020 Jul;86(7):1281-1288. doi: 10.1111/bcp.14193. Epub 2020 May 18. PMID 31823381
- [Background] Richards A. Cardiovascular risk in hypertension: open questions about HOPE 4. Lancet. 2020 Aug 1;396(10247):310. doi: 10.1016/S0140-6736(20)30613-9. No abstract available. PMID 32738948
- [Background] Wagstaff A. Inequality aversion, health inequalities and health achievement. J Health Econ. 2002 Jul;21(4):627-41. doi: 10.1016/s0167-6296(02)00006-1. PMID 12146594
- [Background] Diabetes Project of Department of Public Health. Report on National Survey of Diabetes Mellitius and Risk Factors for Non-communicable Diseases in Myanmar (2014). Myanmar: Myanmar Ministry of Health and Sports, 2014.
- [Background] Naing C, Aung K. Prevalence and risk factors of hypertension in myanmar: a systematic review and meta-analysis. Medicine (Baltimore). 2014 Nov;93(21):e100. doi: 10.1097/MD.0000000000000100. PMID 25380081
- [Background] Zaw KK, Nwe N, Hlaing SS. Prevalence of cardiovascular morbidities in Myanmar. BMC Res Notes. 2017 Feb 15;10(1):99. doi: 10.1186/s13104-017-2422-2. PMID 28202069
- [Background] Bjertness MB, Htet AS, Meyer HE, Htike MM, Zaw KK, Oo WM, Latt TS, Sherpa LY, Bjertness E. Prevalence and determinants of hypertension in Myanmar - a nationwide cross-sectional study. BMC Public Health. 2016 Jul 18;16:590. doi: 10.1186/s12889-016-3275-7. PMID 27430560
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Ansbro E, Issa R, Willis R, Blanchet K, Perel P, Roberts B. Chronic NCD care in crises: A qualitative study of global experts' perspectives on models of care for hypertension and diabetes in humanitarian settings. J Migr Health. 2022 Mar 24;5:100094. doi: 10.1016/j.jmh.2022.100094. eCollection 2022. PMID 35434681
- [Background] Jaung MS, Willis R, Sharma P, Aebischer Perone S, Frederiksen S, Truppa C, Roberts B, Perel P, Blanchet K, Ansbro E. Models of care for patients with hypertension and diabetes in humanitarian crises: a systematic review. Health Policy Plan. 2021 May 17;36(4):509-532. doi: 10.1093/heapol/czab007. PMID 33693657
- [Background] Ansbro E, Homan T, Qasem J, Bil K, Rasoul Tarawneh M, Roberts B, Perel P, Jobanputra K. MSF experiences of providing multidisciplinary primary level NCD care for Syrian refugees and the host population in Jordan: an implementation study guided by the RE-AIM framework. BMC Health Serv Res. 2021 Apr 26;21(1):381. doi: 10.1186/s12913-021-06333-3. PMID 33896418
- [Background] Ruby A, Knight A, Perel P, Blanchet K, Roberts B. The Effectiveness of Interventions for Non-Communicable Diseases in Humanitarian Crises: A Systematic Review. PLoS One. 2015 Sep 25;10(9):e0138303. doi: 10.1371/journal.pone.0138303. eCollection 2015. PMID 26406317
- [Background] Wagstaff A. The bounds of the concentration index when the variable of interest is binary, with an application to immunization inequality. Health Econ. 2005 Apr;14(4):429-32. doi: 10.1002/hec.953. PMID 15495147
- [Background] Tiberti M, Costa V. Disability Measurement in Household Surveys : A Guidebook for Designing Household Survey Questionnaires (English) Washington, D.C.: World Bank Group, 2020.